CLINICAL TRIAL: NCT04938050
Title: Diagnostic Accuracy of a Specialized Pro Forma in Assessing Morbidly Adherent Placenta With Correlation to Intra-operative Findings
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Fatma Fathy Hafez Ismail, Principle investigator, Cairo University
Other Study IDs: 23-2021
Record Dates: First submitted 2021-06-18; First posted 2021-06-24 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Morbidly Adherent Placenta
MeSH Terms: conditions — Placenta Accreta | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasound — Ultrasound evaluation, with grayscale and color Doppler imaging.

SUMMARY:
This study objective is to assess the accuracy of a specialized pro forma in suggesting the probability of Morbidly Adherent Placenta, its extent and its correlation with intraoperative findings.

ELIGIBILITY:
Inclusion Criteria:

* Age group 28:42 years.
* Pregnant women in their late third trimester (34 0/7 weeks: 37 0/7 weeks).
* With a single living fetus in the current pregnancy.
* A previous delivery by at least 1 cesarean section or history of uterine surgery including (surgical evacuation, myomectomy or endometrium ablation)
* Having an anterior placenta previa or anterior low-lying placenta by ultrasound assessment.

Exclusion Criteria:

* Cases with a non-previa placenta, posterior low lying placenta or posterior previa placenta.
* Maternal chronic medical disorders( diabetes mellitus, hypertension)
* Patients presented with severe attack of bleeding.
* Patients presented with rupture of membrane.
* Emergency delivery regardless the cause.

Ages: 28 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 21 pregnant females during their late 3rd trimester between (34 0/7: 37 0/7 weeks gestation)
Sampling Method: Non-Probability Sample
Enrollment: 21 (Estimated)
Dates: Start 2021-06-18 (Actual); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Clinical significance of ultrasound signs in morbidly adherent placenta(most sensitive US sign) | June 2021- July 2022
Accuracy of our specialized pro forma in assessing extent of morbidly adherent placenta(focal , diffuse) | June 2021- July 2022
Accuracy of our specialized pro forma in assessing depth of invasion of placenta accreta spectrum (accrete, increta and percreta) | June 2021- July 2022

SECONDARY OUTCOMES:
1- Correlation between US signs and intraoperative findings including morbidity and mortality | June 2021- July 2022

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university Kasr Alainy OBGYN hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided